CLINICAL TRIAL: NCT07253415
Title: Effects of Adding Thoracic Spine Exercises to Routine Soccer Training on Spinal Alignment and Mobility in Professional Male Soccer Players: a Randomized Controlled Study
Brief Title: Effects of Thoracic Spine Exercises on Spinal Alignment and Mobility in Male Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Kazım Bayram, Lecturer, PhD, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IKCU-FTR-KB-01
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spinal Mobility; Thoracic Spine
Keywords: exercise; thoracic spine; sports; soccer
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The exercise group performed the thoracic spine exercise program in addition to their routine soccer training, while the control group received no intervention and continued their routine training without additional exercises
Who Masked: Outcomes Assessor
Masking Description: The assessor who conducted the outcome measurements was blinded to group allocation. Additionally, all statistical analyses were performed by a biostatistician who was blinded to the study aims.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Players in the exercise group performed thoracic spine exercises in addition to their routine soccer training, three days a week for six weeks, with each session lasting approximately 30-40 minutes. The exercise program comprised six exercises targeting mobility, strength, motor control, and stability of the thoracic region, including thoracic spine extension exercise with foam roller and thoracic extension flexibility exercise, thoracic spine rotation exercise and thoracic rotation exercise in quadrupedal position, open book exercise, and bird-dog exercise. Exercise progression was achieved by systematically increasing repetitions and sets according to the principle of gradual overload and by advancing resistance levels over time.
  Interventions: Other: Thoracic spine exercise
- Control Group (No Intervention): The control group received no intervention and continued their routine training without additional exercises

INTERVENTIONS:
Other: Thoracic spine exercise — Following baseline evaluations, players in the exercise group performed thoracic spine exercises in addition to their routine soccer training, three days a week for six weeks, with each session lasting approximately 30-40 minutes. All players also regularly participated in the routine training program planned by the club technical team, implemented 5 to 6 days a week and lasting approximately 90-120 minutes per session. The exercise program comprised six exercises targeting mobility, strength, motor control, and stability of the thoracic region, including thoracic spine extension exercise with foam roller and thoracic extension flexibility exercise, thoracic spine rotation exercise and thoracic rotation exercise in quadrupedal position, open book exercise, and bird-dog exercise. Exercise progression was achieved by systematically increasing repetitions and sets according to the principle of gradual overload and by advancing resistance levels over time.
  Arms: Exercise Group

SUMMARY:
Thoracic spine mobility is essential for trunk stability, rotational movement, and athletic performance in soccer players. This study aimed to investigate the effects of adding thoracic spine exercises to routine soccer training on spinal alignment, segmental mobility, and thoracic rotation in professional male players.

DETAILED DESCRIPTION:
Soccer is a dynamic and multifaceted sport that involves complex movement patterns, including high-speed running, sudden stops and changes of direction, jumping, collisions, and trunk rotation. The spine serves not only as a central component of the skeletal system but also as a dynamic structure essential for trunk stability, postural control, balance, and efficient force transmission. In athletes, maintaining coordination between body segments, ensuring efficient functioning of the kinetic chain, and sustaining high-level motor control all require optimal spinal function. In high-contact and high-intensity sports such as soccer, the spine is exposed to substantial repetitive loads due to its anatomical structure, which can result in microstructural stress accumulation, postural deviations, and segmental dysfunctions over time, ultimately reducing performance and increasing the risk of injury.

A review of the current literature shows that interventions for trunk control and spinal health in soccer players predominantly focus on the core and lumbar regions, while exercises targeting the thoracic region are not systematically addressed.

Research on spinal exercise interventions and their effects on spinal structure, segmental ROM, and functional mobility has been expanding and gaining clinical relevance. Exercise approaches specifically targeting the thoracic region have been shown to support spinal segmental integrity and improve mobility in both the sagittal and frontal planes.

In recent years, thoracic region-specific exercise approaches have been shown to improve postural control as well as upper and lower extremity performance. However, there are limited studies in the current literature directly examining the effects of thoracic exercises on spinal alignment and mobility.

The present study aimed to examine and compare the effects of a 6-week thoracic spine exercise program on spinal alignment and mobility in professional male soccer players. We hypothesized that 6 weeks of thoracic spine exercises would improve spinal alignment and mobility and that significant differences would be observed between the exercise and control groups in this population.

Forty-nine professional male soccer players from a Second League soccer club were assessed for eligibility. Inclusion criteria were voluntary participation and regular attendance at team training sessions. Exclusion criteria included a history of major sports injuries requiring surgery or injuries that caused time loss, musculoskeletal deformities of the lower and upper extremities, a history of injury within the last 3 months, and spinal trauma within the last 6 months. A total of five players were excluded from the study for not meeting the inclusion criteria. Following baseline assessments, the remaining 44 players were randomly assigned to the exercise group (n = 22) or control group (n = 22). During the study, two players from each group were lost to follow-up, resulting in a final sample of 21 players per group.

Participants were randomly assigned to groups using a computer-generated random sequence (simple randomization). The assessor who conducted the outcome measurements was blinded to group allocation. Additionally, all statistical analyses were performed by a biostatistician who was blinded to the study aims.

All players were provided with detailed information regarding the nature and scope of the study, potential risks, and anticipated benefits prior to participation. Informed consent was obtained from each player before enrollment. The study was conducted in accordance with the Declaration of Helsinki.

All players participated in a detailed information session outlining the interventions and assessment procedures. Assessments were conducted before (pre-test) and after (post-test) the 6-week intervention period. The exercise group performed the thoracic spine exercise program in addition to their routine soccer training, while the control group received no intervention and continued their routine training without additional exercises.

Following baseline evaluations, players in the exercise group performed thoracic spine exercises in addition to their routine soccer training, three days a week for six weeks, with each session lasting approximately 30-40 minutes.

Spinal alignment and mobility of the players were assessed using the Valedo®Shape device (Idiag, Fehraltorf, Switzerland).

An iPhone (Apple Inc., Cupertino, CA, USA) and the Compass application were used to measure thoracic rotation.

All statistical analyses were conducted using IBM SPSS Statistics, Version 26 (IBM., Armonk, NY). Descriptive data are presented as mean ± standard deviation (SD). The normality of data distribution was assessed using the Shapiro-Wilk test. Pre-test differences between the exercise and control groups for all variables were evaluated using one-way ANOVA, and homogeneity of variances was confirmed using Levene's test. Two-way repeated-measures ANOVA was used to analyze main effects and interactions for all variables. Effect sizes were interpreted as small (ηp² < 0.01), medium (ηp² = 0.02-0.1), and large (ηp² > 0.1) [41,42]. When significant main or interaction effects were observed, post-hoc analyses were performed using paired t-tests with Bonferroni correction to determine differences between pre-test and post-test values within each group. Within-group effect sizes (Cohen's d) were calculated as d = (M1 - M2)/σpooled, with values of 0.00-0.19 considered negligible, 0.20-0.49 small, 0.50-0.79 medium, and ≥ 0.80 large. The significance level (α) was set at 0.05.

Thoracic spine exercises, when added to routine training, were found to positively affect spinal alignment and mobility in professional male soccer players. Specifically, they increased lumbar and sacral angles, thoracic, lumbar, sacral, and inclination mobility in the sagittal plane, and bilateral thoracic rotation angles.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who voluntarily agree to participate in the study
* Individuals who regularly attend team training sessions within their club

Exclusion Criteria:

* Individuals who have experienced any sports-related injury within the past 3 months.
* Individuals with conditions that may negatively affect balance or coordination.
* Individuals with musculoskeletal deformities affecting the upper or lower extremities.
* Individuals participating in training programs outside of regular team practices.
* Individuals with a history of spinal surgery, spinal root compression, thoracic pain or tenderness, spinal cord tumors, or spinal trauma.
* Individuals who have experienced trauma to the spinal region within the past 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Spinal Alignment and Mobility Evaluation | six weeks
  Spinal alignment and mobility of the players were assessed using the Valedo®Shape device (Idiag, Fehraltorf, Switzerland). This device evaluates posture and mobility of the thoracic (T1-T2 to T11-T12) and lumbar (T12-L1 to the sacrum) spine in the sagittal and frontal planes. The Valedo®Shape is a non-invasive, computer-assisted measurement system that provides valid and reliable results comparable to radiographic analysis and does not involve radiation exposure. The spinous processes of the spine were marked as anatomical reference points. The Valedo®Shape device was then moved downward by the assessor along all spinous processes, beginning from the C7 vertebra to approximately the S3 level. For the sagittal plane evaluation, measurements were obtained in three positions: neutral posture, maximum flexion, and maximum extension. For the frontal plane evaluation, measurements were taken in the neutral posture as well as during right and left lateral flexion.

SECONDARY OUTCOMES:
Evaluation of Thoracic Rotation | six weeks
  An iPhone (Apple Inc., Cupertino, CA, USA) and the Compass application were used to measure thoracic rotation. Players were asked to sit, cross their hands in front of their chest, and hold a stick between their arms at shoulder height. The phone was placed at the T1-T2 level, and the measurement started from the position from the 0° position. While maintaining contact with the phone, players performed active thoracic rotation, and the resulting angular value was recorded. Players were then asked to return to 0°, and the test was concluded. This method has been reported to demonstrate high reliability (ICC: 0.87). Measurements were repeated three times, and the average value was included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Bayram, Ph.D, Principal Investigator — Izmir University of Economics
Locations (1):
- Altınordu Football Club - Metin Oktay Training Facilities, Izmir, Torbalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves only professional football players and is conducted at a single center.